CLINICAL TRIAL: NCT05989321
Title: A New Approach for Catheter Ablation of Atrial Fibrillation: a Retrospective Cohort Study
Brief Title: A New Approach for Catheter Ablation of Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, mingli Zhou, associate chief physician, The Second Affiliated Hospital of Kunming Medical University
Other Study IDs: IIT-2023-0052-XXG-004
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PVI alone group: Patients who undergo PVI alone using ThermoCool SmartTouch catheter.
  Interventions: Procedure: PVI alone
- PVI + SPs ablation group: Patients who undergo PVI + SPs ablation using ThermoCool SmartTouch catheter.
  Interventions: Procedure: PVI + SPs ablation

INTERVENTIONS:
Procedure: PVI alone — pulmonary vein isolation
  Groups: PVI alone group
Procedure: PVI + SPs ablation — pulmonary vein isolation + SPs ablation
  Groups: PVI + SPs ablation group

SUMMARY:
This is a retrospective cohort study of radiofrequency ablation for the treatment atrial fibrillation(AF). Based on the electrophysiological phenomena found in these cases, the investigators propose a hypothesis regarding the underlying electrophysiological mechanism of AF, as well as a novel approach for catheter ablation of AF.

DETAILED DESCRIPTION:
The investigators propose a new electrophysiological mechanism for AF: the superposition hypothesis. The investigators tested this hypothesis by conducting the retrospective cohort study to determine if superposition potentials (SP) can identify the critical regions where AF is sustained and if ablating SPs can improves the long-term efﬁcacy.

The study consecutively collected patients with underwent the first catheter ablation for symptomatic AF in a university hospital from March 2021 to June 2022, including paroxysmal AF (lasting <7 days), persistent AF (lasting >7 days and <1 year without electrical cardioversion) and long-term persistent AF (lasting >1 year), aged between 18 and 80 years old. AF recurrence was evaluated at 3, 6, 9, and 12 months using 72-hour Holter monitoring at each clinic visit. The eligible patients were divided into two groups: the pulmonary vein isolation(PVI) alone group (n=56) and the PVI + SPs ablation group(n=60).Comprehensive clinical history and procedural data of patients were collected from electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* patients with underwent the first catheter ablation for symptomatic AF

Exclusion Criteria:

* patients with more than one missing follow-up would be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These cases are from a university hospital
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
freedom from AF within 12 months | 12 months
  AF recurrence was evaluated at 3, 6, 9, and 12 months using 72-hour Holter monitoring at each clinic visit. AF recurrence was defined as the occurrence of AF lasting at least 30 seconds after the 3-month blanking period.

SECONDARY OUTCOMES:
the acute termination of AF during the procedure | during the procedure
  Conversion of AF to normal sinus rhythm or atrial tachyarrhythmias during ablation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mingli Zhou, M.D., Principal Investigator — The Second Affiliated Hospital of Kunming Medical University
Locations (1):
- The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505